CLINICAL TRIAL: NCT03725969
Title: The Effect of Camel Milk on Insulin and Incretin Response to a Mixed-meal Challenge in People With Normal Glucose Tolerance
Brief Title: Effect of Camel Milk on Insulin and Incretin Response
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Imperial College London Diabetes Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Other
Other Study IDs: IREC033
Record Dates: First submitted 2018-10-14; First posted 2018-10-31 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Insulin Sensitivity; Glucose Tolerance
MeSH Terms: conditions — Insulin Resistance | interventions — Milk

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy individuals (camel milk) (Experimental)
  Interventions: Dietary Supplement: Camel milk
- Healthy individuals (cow milk) (Experimental)
  Interventions: Dietary Supplement: Cow milk

INTERVENTIONS:
Dietary Supplement: Camel milk — Camel Milk administered 10 minutes before a mixed meal of carbohydrate and protein; 2-week washout between interventions
  Arms: Healthy individuals (camel milk)
Dietary Supplement: Cow milk — Cow milk administered 10 minutes before a mixed meal of carbohydrate and protein;2-week washout between interventions
  Arms: Healthy individuals (cow milk)

SUMMARY:
To examine the differential effect of camel and cow milk on the physiological response, to a liquid mixed-meal challenge, in people with normal glucose tolerance

DETAILED DESCRIPTION:
Camel milk is used as a traditional remedy throughout the Middle East and Indian Subcontinent for conditions such as type 2 diabetes and dyslipidemia. It is currently unclear how such an effect could be mediated in vivo and studies are limited. We performed this study as a pilot experiment to assess the effects of camel milk on Insulin, Glucose, GLP-1, C-peptide and Lipid profile.

ELIGIBILITY:
Inclusion Criteria:

* Normal glucose tolerance
* BMI < 30 kg/m2

Exclusion Criteria:

* Type 1 diabetes mellitus
* Type 2 diabetes mellitus
* Impaired fasting glucose or impaired glucose tolerance
* Lactose intolerance
* Weight loss / gain ≥ 5 kg in the preceding two months
* Use of estrogenic drugs or corticosteroids
* Known hypertriglyceridemia requiring treatment
* History of heart attack, angina or cardiovascular disorder
* History of malignant tumor
* Pregnant or lactating women
* Hemoglobin < 12 for any reason
* Recent surgery or major hemorrhage
* History of bariatric or metabolic surgery

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2017-02-01 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Glucose response to camel and cow milk | 5 months
  The difference between interventions in terms of peak of glucose
Response of glucose to camel and cow milk | 5 months
  The difference between interventions in terms of area under the curve

SECONDARY OUTCOMES:
Insulin response to camel and cow milk | 5 months
  The difference between interventions in terms of peak
Response of insulin to camel and cow milk | 5 months
  The difference between interventions in terms of area under the curve
GLP-1 response to camel and cow milk | 5 months
  The difference between interventions in terms of peak
Response of GLP-1 to camel and cow milk | 5 months
  The difference between interventions in terms of area under the curve
C-peptide response to camel and cow milk | 5 months
  The difference between interventions in terms of peak
Response of C-peptide to camel and cow milk | 5 months
  The difference between interventions in terms of area under the curve

CONTACTS AND LOCATIONS:
Overall Officials: Dr Nader Lessan, MBBS MD FRCP, Principal Investigator — Imperial College London Diabetes Centre
Locations (1):
- Imperial College London Diabetes Centre, Abu Dhabi, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No